CLINICAL TRIAL: NCT05548725
Title: Relation Between Acute Kidney Injury and Mineral Bone Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Asmaa Ahmed Mohamed Abd Elraheem, Director, Assiut University
Other Study IDs: Relation between AKI and BMD
Record Dates: First submitted 2022-09-11; First posted 2022-09-21 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Reguired field — Investigations to know relationship between acute kidney injury and mineral bone disease

SUMMARY:
Relation between acute kidney injury and mineral bone disease

DETAILED DESCRIPTION:
Assiut Medical School Research Proposal Form 2 Part 2: Research Details 2.1 Background (Research Question, Available Data from the literature, Current strategy for dealing with the problem, Rationale of the research that paves the way to the aim(s) of the work).

Numerous studies have evaluated the prevalence and importance of mineral and bone disorders among patients with chronic kidney disease (CKD) and end-stage renal disease (ESRD). However, little is known about dysregulated mineral and bone metabolism in acute kidney injury (AKI) [ Acute kidney injury is the new consensus term for acute renal failure It refers to a clinical syndrome characterised by a rapid (hours to days) decrease in renal excretory function, with the accumulation of products of nitrogen metabolism such as creatinine and urea and other clinically unmeasured waste products. Other common clinical and laboratory manifestations include decreased urine output (not always present), accumulation of metabolic acids, and increased potassium and phosphate concentrations. The term acute kidney injury has replaced acute renal failure to emphasise that a continuum of kidney injury exists that begins long before sufficient loss of excretory kidney function can be measured with standard laboratory tests. The term also suggests a continuum of prognosis, with increasing mortality associated with even small rises in serum creatinine, and additional increases in mortality as creatinine concentration rises. The incidence of acute kidney injury (AKI) is increasing among hospitalized patients . Treating the condition consumes significant amounts of resources even after hospital discharge

. Although AKI was once considered a reversible condition, mounting evidence has indicated that AKI may have a negative impact upon subsequent renal function and long-term prognosis, even if kidney

ELIGIBILITY:
Inclusion Criteria:

* 200 patients with acute kidney injury and their relationship to mineral bone disease.

Exclusion Criteria:

* Non hypertensive
* Non cardiac
* Active malignancy
* Acute or chronic liver disease
* Acute poisoning
* Covid

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: c. Sample Size Calculation: 200 cases , 200 controls from December 2021to December 2023 2.4.4 -Study tools (in detail, e.g., lab methods, instruments, steps, chemicals, …):
  Study techniques:
  a) Full (thorough) history & clinical examination. b) Laboratory investigations:
  * Blood Urea, Serum creatinine
  * Pth
  * Ph
  * Ca
  * Na
  * k
  * Mg
  * Vit d
  * Other routine investigations c) Imaging:
  * Abdominal U/S d) ECG 2.4.5 -Research outcome measures:
    a. Primary (main):
  * Identify the association between Acut
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-09-25 (Estimated); Primary Completion 2023-09-25 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Relation between AKI and mineral bone disease | Baseline
  Relationship between acute kidney injury and mineral bone disease

REFERENCES:
- [Background] Agar A, Gulabi D, Sahin A, Gunes O, Hancerli CO, Kilic B, Erturk C. Acute kidney injury after hip fracture surgery in patients over 80 years of age. Arch Orthop Trauma Surg. 2022 Sep;142(9):2245-2252. doi: 10.1007/s00402-021-03969-y. Epub 2021 May 31. PMID 34056678
- [Background] Koizumi M, Komaba H, Fukagawa M. Parathyroid function in chronic kidney disease: role of FGF23-Klotho axis. Contrib Nephrol. 2013;180:110-23. doi: 10.1159/000346791. Epub 2013 May 3. PMID 23652554
- [Result] Wesseling-Perry K, Salusky IB. Phosphate binders, vitamin D and calcimimetics in the management of chronic kidney disease-mineral bone disorders (CKD-MBD) in children. Pediatr Nephrol. 2013 Apr;28(4):617-25. doi: 10.1007/s00467-012-2381-8. Epub 2013 Feb 5. PMID 23381010